CLINICAL TRIAL: NCT03059758
Title: Deductive Reasoning and Math Learning Difficulty: an fMRI Study in Children
Brief Title: Deductive Reasoning and Math Learning Difficulty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0686
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brain activity during reasoning and measure of math skill (Experimental): Brain activity during reasoning and measure of math skill
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI — All participants are scanned while evaluating deductive reasoning problems. Their math skill is also assessed.
  Other Names: fMRI scanning

SUMMARY:
Most studies to date that have examined the factors underlying math achievement in children have focused on basic numerical knowledge. Yet, math skills are clearly not limited to basic numerical knowledge and recent behavioral studies suggest a relationship between math and deductive reasoning skills. The goal of this study is to determine the neural mediators of this relationship using functional magnetic resonance imaging. The investigators will ask children from 8 to 14 to complete a standardized math achievement test, and measure their brain activity while they process deductive arguments. The investigators will then correlate brain activity during reasoning to individual math skills to identify the brain regions in which activity during reasoning is modulated by math skill.

ELIGIBILITY:
Inclusion Criteria:

* Girl or boy between 8 and 14
* Right-handed
* Affiliated to the French social security
* Whose parents gave informed consent

Exclusion Criteria:

* Neurological disorders
* Psychiatric disorders
* Birth complications requiring admission into neonatal intensive care unit
* Medication affecting central nervous system processing
* Significant hearing impairment
* Uncorrected visual impairment
* Non-native French speaker
* Contraindications for MRI

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 137 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Correlation between brain activity during deductive reasoning and math skill 18 to 24 months later | 18 to 24 months after scanning
  Brain activity measured using fMRI and math skill measured using a standardized test 18 to 24 months after scanning

CONTACTS AND LOCATIONS:
Locations (1):
- CH le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwartz F, Epinat-Duclos J, Leone J, Poisson A, Prado J. Neural representations of transitive relations predict current and future math calculation skills in children. Neuropsychologia. 2020 Apr;141:107410. doi: 10.1016/j.neuropsychologia.2020.107410. Epub 2020 Feb 22. PMID 32097661